CLINICAL TRIAL: NCT00931242
Title: A Phase 2, Open-label, Investigator-Initiated Study to Evaluate the Safety and Efficacy of Apremilast in Subjects With Recalcitrant Contact or Atopic Dermatitis
Brief Title: Study of Apremilast in Atopic or Contact Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Alice B. Gottlieb, MD, PhD, Tufts Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD / CD; AP-ECZ-PI-0030 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2009-06-30; First posted 2009-07-02 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-11

CONDITIONS: Atopic Dermatitis; Allergic Contact Dermatitis
Keywords: eczema; dermatitis; TNF blockade; PDE4 inhibitor; T cell inhibitor
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis, Allergic Contact; Eczema; Dermatitis | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Apremilast (Experimental): Apremilast is being evaluated at daily doses of 20 mg by mouth (PO) twice daily (BID) for 12 weeks of treatment (treatment phase) in subjects with recalcitrant plaque-type Atopic Dermatitis (AD) or Allergic Contact Ddermatitis (ACD).
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast is being evaluated at daily doses of 20 mg by mouth (PO) twice daily (BID) for 12 weeks of treatment (treatment phase) in subjects with recalcitrant plaque-type Atopic Dermatitis (AD) or Allergic Contact Ddermatitis (ACD).
  Other Names: CC-10004 (apremilast)

SUMMARY:
The objective of this study is to evaluate the efficacy of apremilast in patients with recalcitrant atopic or contact dermatitis.

DETAILED DESCRIPTION:
Atopic Dermatitis (AD) is a chronic, inflammatory skin disease characterized by dry, red, and itchy patches that can become thickened and lichenified with time. Contact Dermatitis, or Allergic Contact Dermatitis (ACD), is an eczematous reaction in response to an environmental allergen.

The etiology of Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD) has not been completely elucidated, and new understandings of underlying mechanisms have expanded and focused treatment regimens and paradigms.

Atopic Dermatitis (AD) is thought to be mediated by Th2 type T cells elaborating a number of cytokines which are blocked in vitro by apremilast. The chronic Atopic Dermatitis (AD) pathway may involve a change to Th1 cytokines. Genetic factors do not contribute as much to the course of Allergic Contact Dermatitis (ACD) as in Atopic Dermatitis (AD). Rather, Allergic Contact Dermatitis (ACD) is a type IV, T-cell mediated, delayed-hypersensitivity reaction that can be self-limited. Similar to Atopic Dermatitis (AD), a number of pro-inflammatory cytokines are involved in recruiting T cells preferentially to the skin: Th1 cytokines, Th2 cytokines, CD8 cytokines, and T-regulatory cytokines. These pathways in Allergic Contact Dermatitis (ACD) are activated by IFN-γ, driven by TNF-α, and as above, apremilast has been shown to block these cytokines in vitro.

Current treatments for Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD) include skin care, trigger avoidance (especially in the case of ACD), topical corticosteroids, steroid sparing treatments, antihistamines, topical and systemic antibiotics, and ultraviolet light. For more recalcitrant Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD)cases, several immunosuppressive treatments exist.

Subjects with recalcitrant Atopic Dermatitis (AD) or Allergic Contact Dermatitis (ACD)have exhausted conventional systemic treatment options because they do not respond to conventional systemic therapy or cannot use these agents due to side effects or cumulative toxicity.

There is an urgent need to evaluate new therapeutic options in recalcitrant Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD). Very few of the available drugs for recalcitrant Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD) have reasonable efficacy and safety profiles in this condition, are easily available, or easy to administer. A new treatment strategy is needed for the treatment of recalcitrant contact or atopic dermatitis that would increase efficacy, minimize toxicity for both short and long-term treatment, and be easy to administer. The availability of alternative drug treatment(s) offering safe and effective short and long-term management would significantly benefit subjects with recalcitrant contact or atopic dermatitis.

This study uses a novel oral agent (apremilast) that modulates multiple anti-inflammatory pathways through targeted phosphodiesterase type IV (PDE4) inhibition decreased expression of dermatitis. Apremilast has pharmacodynamic properties with a potential therapeutic benefit for treating inflammatory autoimmune disorders that involve elevated serum cytokine levels, including Atopic Dermatitis (AD) and Allergic Contact Dermatitis (ACD).

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign an informed consent form.
* Must be male or female and aged ≥ 18 years at time of consent.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Must have a documented history of contact or atopic dermatitis for at least 3 months prior to screening visit. Subjects will be asked to bring records at the time of screening visit; if they do not bring these records, subjects will be asked to complete and sign a release of records for which will be sent to the subject's physician. The Investigators will review records to confirm eligibility prior to enrolling a subject into the study.
* Subjects must fulfill criteria outlined in at least one of the following clinical categories:

  * Unresponsive to standard systemic or topical therapy, as defined by clinical history, in the investigator's opinion, i.e. inadequate response to one or more adequate treatment course (s) of standard systemic therapy including but not limited to: topical steroids, ultraviolet light A [UVA], narrowband ultraviolet B (NBUVB), ultraviolet light B [UVB].
  * Intolerant to or cannot receive (e.g., contraindication to prescribe) standard systemic or topical therapy for contact or atopic dermatitis.
* Must have a IGA score of at least moderate (3 on a 0 to 5 point scale) at screening.
* Must meet the following laboratory criteria:

  * White blood cell count ≥ 3000/ μL (3 x 109/L) and < 14,000/ μL (< 14 x 109/L)
  * Platelet count > 100,000/ μL (100 x 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * AST (SGOT) and ALT (SGPT) ≤ 1.5 x upper limit of normal (ULN)
  * Hemoglobin > 9 g/dL
  * Total bilirubin ≤ 2.0 mg/dL
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at screening. In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication:

  * oral, injectable, or implantable hormonal contraceptives;
  * tubal ligation;
  * intrauterine device;
  * barrier contraceptive with spermicide;
  * vasectomized partner while on study.
* A FCBP must agree to have pregnancy tests every 4 weeks while on study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in sexual activity with FCBP while on study medication and for 84 days after taking the last dose of study medication.

Exclusion Criteria:

* Inability to provide voluntary consent.
* History of clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic, or other major disease. Potential subjects with severe uncontrolled conditions, such as severe uncontrolled diabetes, will be excluded.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Pregnant or breastfeeding.
* Systemic fungal infection.
* History of active mycobacterial infection with any species (including Mycobacterium tuberculosis) within 3 years prior to screening visit. Subjects with Mycobacterium tuberculosis infection more than 3 years prior to screening visit are allowed if successful treatment was completed at least 3 years prior to randomization and is documented and available for verification.
* Latent Mycobacterium tuberculosis infection as indicated by a positive Purified Protein Derivative [PPD] skin test. Subjects with a positive PPD skin test and documented completion of treatment for latent TB are eligible. Subjects with a positive PPD skin test and not treated or no documentation of completion of treatment are ineligible.
* If QuantiFERON® test is performed instead of the PPD test, only those with a negative QuantiFERON® test are allowed in the study.
* History of incompletely treated Mycobacterium tuberculosis infection as indicated by:

  * Subject's medical records documenting incomplete treatment for Mycobacterium tuberculosis.
  * Subject's self-reported history of incomplete treatment for Mycobacterium tuberculosis.
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years).
* Clinically significant abnormality on the chest x-ray (CXR) at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Contact or atopic Dermatitis flare within 30 days of screening, defined as a sudden intensification of contact or atopic dermatitis
* Use of systemic therapy for contact or atopic dermatitis (including but not limited to cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, tacrolimus, azathioprine) within 14 days of Week 0 (Baseline).
* Topical therapy (including but not limited to topical steroids, topical vitamin A or D analog preparations, tacrolimus, pimecrolimus, or anthralin) within 7 days of Week 0 (Baseline). (Exception: Class VI or VII potency corticosteroids will be allowed [Appendix 18.8] for treatment of the palms, face, scalp, axillae, plantar surfaces and groin in accordance with the manufacturers suggested usage, except within 24 hours of a study visit. Non-medicated emollients [e.g., Eucerin®], and tar shampoo are also allowed.)
* Adalimumab, etanercept, efalizumab or infliximab use within 56 days of Week 0 (Baseline).
* Alefacept use within 180 days of Week 0 (Baseline).
* Phototherapy (PUVA, UVA,NB-UVB, UVB) within 14 days of Week 0 (Baseline).
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer).
* Any clinically significant abnormality on 12-lead ECG at screening.
* History of congenital or acquired immunodeficiency (e.g., Common Variable Immunodeficiency [CVID]).
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening.
* History of Human Immunodeficiency Virus (HIV) infection.
* Antibodies to Hepatitis C at screening.
* Malignancy or history of malignancy (except for treated [i.e., cured] basal-cell skin carcinoma(s) or treated squamous-cell skin carcinomas).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice B. Gottlieb, M.D., PhD., Principal Investigator — Tufts Medical Center, Department of Dermatology
Locations (1):
- Tufts Medical Center, Department of Dermatology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Leung DY, Boguniewicz M, Howell MD, Nomura I, Hamid QA. New insights into atopic dermatitis. J Clin Invest. 2004 Mar;113(5):651-7. doi: 10.1172/JCI21060. PMID 14991059
- [Background] Novak N, Bieber T, Leung DY. Immune mechanisms leading to atopic dermatitis. J Allergy Clin Immunol. 2003 Dec;112(6 Suppl):S128-39. doi: 10.1016/j.jaci.2003.09.032. PMID 14657843
- [Background] Girolomoni G, Sebastiani S, Albanesi C, Cavani A. T-cell subpopulations in the development of atopic and contact allergy. Curr Opin Immunol. 2001 Dec;13(6):733-7. doi: 10.1016/s0952-7915(01)00287-4. PMID 11677098
- [Background] Cavani A, Albanesi C, Traidl C, Sebastiani S, Girolomoni G. Effector and regulatory T cells in allergic contact dermatitis. Trends Immunol. 2001 Mar;22(3):118-20. doi: 10.1016/s1471-4906(00)01815-9. PMID 11286716
- [Background] Cone RE, Li X, Sharafieh R, O'Rourke J, Vella AT. The suppression of delayed-type hypersensitivity by CD8+ regulatory T cells requires interferon-gamma. Immunology. 2007 Jan;120(1):112-9. doi: 10.1111/j.1365-2567.2006.02486.x. Epub 2006 Oct 18. PMID 17052246
- [Background] Jung T, Stingl G. Atopic dermatitis: therapeutic concepts evolving from new pathophysiologic insights. J Allergy Clin Immunol. 2008 Dec;122(6):1074-81. doi: 10.1016/j.jaci.2008.09.042. Epub 2008 Nov 6. PMID 18992925
- [Background] Belloni B, Andres C, Ollert M, Ring J, Mempel M. Novel immunological approaches in the treatment of atopic eczema. Curr Opin Allergy Clin Immunol. 2008 Oct;8(5):423-7. doi: 10.1097/ACI.0b013e32830fb8fd. PMID 18769195
- [Background] Harada D, Takada C, Nosaka Y, Takashima Y, Kobayashi K, Takaba K, Manabe H. Effect of orally administered KF66490, a phosphodiesterase 4 inhibitor, on dermatitis in mouse models. Int Immunopharmacol. 2009 Jan;9(1):55-62. doi: 10.1016/j.intimp.2008.09.011. Epub 2008 Oct 12. PMID 18854230
- [Background] Schmitt J, Langan S, Williams HC; European Dermato-Epidemiology Network. What are the best outcome measurements for atopic eczema? A systematic review. J Allergy Clin Immunol. 2007 Dec;120(6):1389-98. doi: 10.1016/j.jaci.2007.08.011. Epub 2007 Oct 1. PMID 17910890
- [Background] Gottlieb AB, Strober B, Krueger JG, Rohane P, Zeldis JB, Hu CC, Kipnis C. An open-label, single-arm pilot study in patients with severe plaque-type psoriasis treated with an oral anti-inflammatory agent, apremilast. Curr Med Res Opin. 2008 May;24(5):1529-38. doi: 10.1185/030079908x301866. Epub 2008 Apr 16. PMID 18419879

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast: Apremilast is being evaluated at daily doses of 20 mg PO twice daily (BID) for 12 weeks of treatment (treatment phase) in subjects with recalcitrant plaque-type AD or ACD.
- Screen Failures: Patients who were screened but failed to meet inclusion criteria for the study
Period: Overall Study
Arm/Group | Apremilast | Screen Failures
Started | 10 | 2
Completed | 5 | 0
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Apremilast: Apremilast is being evaluated at daily doses of 20 mg PO (by mouth) twice daily (BID) for 12 weeks of treatment (treatment phase) in subjects with recalcitrant plaque-type atopic dermatitis or allergic contact dermatitis.
- Screen Failures: Subjects that were screened but failed to meet inclusion criteria for the study.
- Total: Total of all reporting groups
Arm/Group | Apremilast | Screen Failures | Total
Number analyzed (Participants) | 10 | 2 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 2 | 10
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 43.3 (14.2442971) | 53.4 (4.5) | 45 (13.0384048)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 5 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving an Improvement (Decrease) in IGA (Investigator Global Assessment) by Two or More Points
Description: Improvement in IGA (Investigator Global Assessment) by two or more points on a five point scale, with 0 being no disease activity and 5 being maximum disease activity, at week 12
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Apremilast
Number analyzed (Participants) | 10
participants | 2

2. Secondary Outcome: Number of Patients Achieving 75% Reduction in Eczema Area and Severity Index (EASI) Score at Week 12 in Reference to Week 0
Description: EASI scores range from 0 to 72, with higher scores reflecting greater disease severity. Erythema, edema, lichenification, and excoriations/erosions are scored on a scale of 0 (none) to 3 (severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 to 6. The total qualitative score is multiplied by the degree of involvement for each anatomic region and then multiplied by a constant and summed to yield the EASI score.
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Apremilast
Number analyzed (Participants) | 10
participants | 1

3. Secondary Outcome: Number of Patients Achieving 50% Reduction in Eczema Area and Severity Index (EASI) Score at Week 12 in Reference to Week 0
Description: as for outcome 2
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Apremilast
Number analyzed (Participants) | 10
participants | 2

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Apremilast
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=12)
Sepsis 2nd to Atopic Dermatitis (Infections and infestations) | 1 (1) — This patient was in the screening phase of the trial and never received study medication. The subject was not eligible to enroll in trial due to the infection and flare of dermatitis.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apremilast (N=12)
Conjunctivitis (Eye disorders) | 1 (1) — routine questioning at visit
Headache (Nervous system disorders) | 2 (2) — routine questioning at visit
Burn (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visit
Nausea (Gastrointestinal disorders) | 2 (2) — routine questioning at visit
asymptomatic sinus arrythmia per EKG (Cardiac disorders) | 1 (1) — routine EKG
GI upset (Gastrointestinal disorders) | 1 (1) — routine questioning at visit
soft stool (Gastrointestinal disorders) | 1 (1) — routine questioning at visit
dermatitis flare (Skin and subcutaneous tissue disorders) | 4 (4) — routine questioning at visit
foot fracture after mechanical fall (Musculoskeletal and connective tissue disorders) | 1 (1)
rigors (Nervous system disorders) | 1 (1) — routine questioning at visit
insomnia (Nervous system disorders) | 1 (1) — routine questioning at visit
seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visit
facial irritation from ketoconazole (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visit
ectropion (Eye disorders) | 1 (1) — routine questioning at visit
flatulence (Gastrointestinal disorders) | 1 (1) — routine questioning at visit
upper respiratory infection (Infections and infestations) | 2 (2) — routine questioning at visit
atopic blepharoconjunctivitis (Eye disorders) | 1 (1) — routine questioning at visit
meibomian gland dysfunction (Eye disorders) | 1 (1) — routine questioning at visits
myalgias (Nervous system disorders) | 1 (1) — routine questioning at visits
chills (Nervous system disorders) | 1 (1) — routine questioning at visits
lower back pain 2nd to motor vehicle accident (minor) (Musculoskeletal and connective tissue disorders) | 1 (1) — routine questioning at visits
b12 deficiency (Blood and lymphatic system disorders) | 1 (1) — pcp screening
increase in number of stools (Gastrointestinal disorders) | 1 (1) — routine questioning at visits
hair dye allergy (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visits
diverticulosis (Gastrointestinal disorders) | 1 (1) — screening colonoscopy
internal hemorrhoids (Gastrointestinal disorders) | 1 (1) — screening colonoscopy
scraped shin from mechanical injury (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visits
nodules in breasts (Skin and subcutaneous tissue disorders) | 1 (1) — physical examination (routine)
MSSA skin infection (Skin and subcutaneous tissue disorders) | 1 (1) — routine questioning at visits

LIMITATIONS AND CAVEATS:
This was a small, single-arm open-label study with no placebo or comparison group to serve as a control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No